## NCT04916444

Title: Dystonia Treatment With Injections Supplemented By Transcranial Magnetic Stimulation

Document Date: 7/21/2024

The primary outcome was the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS). Participant exam was videotaped and the TWSTRS score was determined by two blinded raters who are fellowship-trained movement disorder neurologists. Secondary outcomes included non-motor symptoms such as mood measured by the Beck Depression Inventory (BDI), cognitive tasks measured by the Wisconsin Card Sorting Task (WCST) and Trail Making Tests (TMT A and B), and gait measured by the Zeno walkways system. In addition, patient-reported outcomes were collected regarding adverse events, tolerability, and predictions regarding the active versus the sham coil.

Two-way repeated measures ANOVA was used for statistical analysis of the primary and secondary outcomes. The statistical analyses were performed using SPSS. The Benjamini-Hochberg procedure was applied to control the false discovery rate for multiple comparisons of the secondary outcomes.